CLINICAL TRIAL: NCT02622529
Title: Patients' Conscious Experience and Psychological Consequences of Awake Surgery for Intracerebral Lesions
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Nader Hejrati, med. pract., Cantonal Hospital of St. Gallen
Other Study IDs: EKSG 15/157
Record Dates: First submitted 2015-11-30; First posted 2015-12-04 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Fear; Anxiety; Stress
Keywords: Awake craniotomy; Psychological consequences; Fear and Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening through Questionnaires: All of the patients within this single existent Arm will receive the questionnaires.
  Interventions: Other: Screening through questionnaires

INTERVENTIONS:
Other: Screening through questionnaires — Distribution of Questionnaires to every participant within the single existent Arm at three times.

SUMMARY:
This study aims to investigate patients' experience of awake surgery of the brain. Patients therefore must suffer a disease that makes the technique of awake craniotomy necessary.

In more detail, the investigators are performing this study in order to investigate the influence of fear on pain perception during surgery for patients undergoing awake surgery for lesions within the brain. In the event of finding a correlation between fear of the surgery and intraoperative pain perception, the investigators aim to reduce possible fear beforehand.

An additional goal of the investigators is to identify psychological consequences of awake craniotomy timely and admit patients to an adequate therapy if necessary.

There will be no changes regarding the actual treatment of the disease. In case of a consent, the patient will receive questionnaires at three timepoints: 1. day before surgery. 2. third day after surgery. 3. at 3-6 months postoperatively at the outpatient clinics.

The benefit of participating in this study is the possibility of detecting psychological consequences of awake craniotomy at an early stage. If required, patients will then receive treatment timely.

There are no additional risks. Theoretically there is only a data risk after analysis.

Patients are free to decide if they want to participate within this study. There are no changes in the actual treatment if patients deny participation. In case of participation, patients have the right to quit at any time with no reasoning at all.

During the study investigators are collecting health-related data. If patients quit before the study end, data will still be used in pseudonymized form. After 10 years, data will be destroyed.

In case of participation the only duty for the patient is to fill out the questionnaires at the above mentioned three time points.

The investigators conduct this study based on all rules of law regarding data protection. Investigators only use the collected data in relation to this study. All investigators are under obligation to secrecy.

DETAILED DESCRIPTION:
ETHICAL AND REGULATORY ASPECTS

Ethical Conduct of Study

The research project will be carried out in accordance to the research plan and with principles enunciated in the current version of the Declaration of Helsinki (DoH), the Essentials of Good Epidemiological Practice issued by Public Health Switzerland (EGEP), the Swiss Law and Swiss regulatory authority's requirements as applicable. The EC and regulatory authorities will be informed about project start and termination.

The Project Leader of this Project Leader initiated Trial acknowledges his responsibilities as both the Investigator and the Project Leader.

Risk categorisation

Risk category A: Enroled patients are not exposed to additional risks, as intraoperative mapping of brain functions using electrical stimulation in awake patients is actually considered the gold standard of treatment in intracerebral lesions in the immediate vicinity or within eloquent brain regions.

Ethics Committee (EC)

Before the project will be conducted, the project plan, the proposed participant information and consent form as well as other project-specific documents shall be submitted to a competent Ethics Committee (EC). The regular end, premature end or interruption of the research project is reported to the EC within 90 days upon completion of the project (HRO Art. 22).

Participant Information and Informed Consent

Consecutive ongoing recruitment through investigator(s) in daily clinical practice (consultations). The subjects will receive the consent form with an address and phone number indicated where further questions regarding the study can be discussed directly with the project leader. This will take place at least one week before the hospitalisation.

Participant privacy and safety

The Project Leader affirms and upholds the principle of the participants' right to dignity, privacy and health and that the project team shall comply with applicable privacy laws. Especially, anonymity of the participants shall be guaranteed when presenting the data at scientific meetings or publishing them in scientific journals.

Individual participant medical information obtained as a result of this research project is considered confidential and disclosure to third parties is prohibited. Participant confidentiality will be further ensured by utilising identification code numbers to correspond to medical information in the computer files.

For data verification purposes, authorised representatives of the Project Leader, a competent ethics committee may require direct access to parts of the medical records relevant to the project, including participants' medical history.

Early termination of Project

The Project Leader (and any competent authority) may terminate the project prematurely according to certain circumstances (insufficient participant recruitment, change of project leader or any other reason that would prevent the project execution according to the research plan). The premature end or interruption of the research project would be reported to the EC within 90 days upon completion of the project (HRO Art. 22).

Amendments, Changes

Significant changes to the project plan would be communicated to relevant parties (e.g., investigators, EC). The Project Leader would submit to the EC any application documents, which are affected by the change. At the same time, the project leader would provide information on the reasons for the change. Substantial amendments are only implemented after approval of the EC.

BACKGROUND

Intraoperative mapping of brain functions using electrical stimulation in awake patients has been proven to be a safe technique that enables increased tumor removal while preserving the functional status of the patients. Former studies reported that the conscious experienced procedure is generally well tolerated and psychological sequelae due to awake craniotomy seem to be rare (Milian et al., 2014). Fear, anxiety and pain are the most commonly seen phenomena intraoperatively (Milian et al., 2014). It is also known that fear and anxiety may aggravate pain perception (Keefe et al., 2001). The investigators hypothesize that patients with less preoperative anxiety experience less intraoperative pain.

Rationale for the research Project

Potential postoperative psychological sequelae could be considered and affected patients could benefit of early recognition and treatment.

Risk-Benefit Assessment

Enroled patients are not exposed to additional risks, as intraoperative mapping of brain functions using electrical stimulation in awake patients is actually considered the gold standard of treatment in intracerebral lesions in the immediate vicinity or within eloquent brain regions. Potential postoperative psychological sequelae could be considered and affected patients could benefit of early recognition and treatment.

PROJECT DESIGN

Type of research and general project design

Research project in which health-related personal data is collected. Data will be pseudonymized. Prospective, monocentric, descriptive, cohort study. Overall study duration will be about one year. Patients are recruited at the investigators in daily clinical practice, which can be days to weeks prior to surgery. Once the surgery is started the study duration for each patient will last 6 months post-surgery.

Procedures

Standardized questionnaires will be completed by the selected patients as follows:

1st day preoperatively: MMSE, NRS-anxiety, HADS-D, PDS-1, BPI, PHQ-D, BDI. Intraoperatively: NRS for anxiety and pain at three timepoints during surgery: before skin incision, after removal of the bone flap, after tumor resection.

3rd day postoperatively: HADS-D, PHQ-D, PDS-1, BPI, NRS for pain. 6 months postoperatively at the outpatient clinics: PHQ-D, BDI, HADS-D, PDS-1, BPI.

Recruitment and Screening

Consecutive ongoing recruitment through investigator(s) in daily clinical practice (consultations). The subjects will receive the consent form with an address and phone number indicated where further questions regarding the study can be discussed directly with the project leader. This will take place at least one week before the hospitalisation.

Methods of minimising bias

The use of validated questionnaires. Blinding is not necessary as there are no randomized/different therapies offered. Additional factors to be considered as they influence primary and secondary endpoints: Assessment of gender and age.

STATISTICAL METHODOLOGY

The study is a non-interventional, monocentric cohort study. The scores which will be analysed as primary and secondary endpoints are in general not assumed to follow a normal distribution. Differences in the raw (untransformed) scores and for changes of the scores over time, will be described by descriptive statistics. The hypotheses of the primary and secondary endpoints described below, will not be examined by any statistical tests.

Hypothesis

The investigators hypothesize that intraoperative pain perception, measured by the NRS, in patients with less preoperative fear and anxiety must be lower. The scores listed as secondary endpoints are hypothesized not to change between pre- and post-operative measurement.

As the expected sample size is not large enough to carry out a statistical test with adequate power, no hypothesis testing will be carried out for this study. The evidence for differences in the scores of the primary and secondary endpoints will be discussed based on the descriptive statistics.

Determination of Sample Size

The primary objective of this study is of descriptive nature, i.e., to assess the conscious experience and experience and psychological consequences of awake surgery among the patient collective at the Cantonal Hospital St. Gallen (Kantonsspital St. Gallen, KSSG). The number of included patients is governed by the duration of the study, which is planned to be one year. Within this year it is expected that around 20 patients, recruited at the KSSG, will be included in the study.

Statistical criteria of termination of Trial

There will be no statistical criteria, which would trigger early termination of this trial, as long as the data gathering process is not impaired.

Planned Analyses

The following measures will be reported: mean, standard deviation, 95% confidence interval, median, 1st and 3rd quartile, minimum, and maximum.

Further the same descriptive statistics will be reported for patient characteristics on continuous scale (e.g. age) and percentages will be reported for categorical variables (e.g. gender). The Spearman rank correlation, which is a non-parametric measure for correlations, for the same scores measured at different occasions, will be reported for the scores in the primary and secondary endpoint.

Datasets to be analysed, analysis populations

The analysis population includes all eligible patients which were recruited in the study. Patients will be included in the analysis if they have included any of the questionnaires. Characteristics of patients which did not meet the inclusion criteria will be reported separately. If a patient has a missing value, or missed a follow-up visit, only the observed measurements will be included and no data imputation will be applied. This implies that the data will be analysed according to the intention to treat principle, which should not be problematic as no intervention is planned in this study.

Essentially no subgroup analyses are planned but under the assumption of equal group sizes, a descriptive analysis of the examined scores for subgroups of gender and age will complement the analysis.

Primary Analyses

Descriptive statistics will be displayed for the NRS score and for the changes in the NRS score between the pre-operative and intra-operative and the pre-operative and post-operative measurements.

Secondary Analyses

For the measures of the secondary analysis (PHQ-D, BDI, MMSE, HADS-D, PDS-1 and BPI) descriptive statistics for each measurement occasion and for the changes in the measures will be carried out.

Interim Analyses

No interim analysis is planned. The duration of the study will be one year. However, interim analyses are possible if requested by the investigator, as the data will be analysed with descriptive statistics only and no intervention is planned.

Deviations from the original statistical plan

Deviations from the planned statistical analysis will be documented and justified in the final statistical report.

Handling of missing data and drop-outs

Patients who have not submitted any of the questionnaires will be excluded from the analysis. However, patient characteristics for patients submitting and not or only partially submitting questionnaires will be compared to determine if there are any statistically significant or clinically relevant differences between the two groups. This may affect how the results of the study should be interpreted.

DATA AND QUALITY MANAGEMENT

Data handling and record keeping / archiving

All data will be recorded in an excel-file, only accessible by authorised personnel, such as Werner Surbeck, Hejrati Nader. The questionnaires will be saved by Werner Surbeck in his locked bureau during the study. On the Case Report Forms (CRF) and other project specific documents, subjects are not identified by their names, but by a unique subject number (UPN).

Confidentiality, Data Protection

Project data will be handled with uttermost discretion and is only accessible to authorized personnel who require the data to fulfil their duties. On the CRFs and other project specific documents, subjects are not identified by their names, but by a unique subject number (UPN). UPN will not consist of initials of the subjects or their date of birth.

The UPN will be distributed to all subjects to whom the questionnaires will be given and used from this moment on exclusively. Subject identification list will be compiled and stored by Dr W. Surbeck in an Excel sheet only on his personal laptop secured by a strong password. A regular backup of the subject identification list will be stored on a Universal Serial Bus (USB) device by Dr Surbeck and locked securely in his office. All alterations in the list will be done by Dr W. Surbeck exclusively.

Coding

On the CRFs and other project specific documents, subjects are not identified by their names, but by a unique subject number (UPN).

Archiving and Destruction

All trial data, including documents necessary for patient identification and post-trial care, will be archived for a minimum of 10 years upon premature- or trial termination.

ANNNOUNCEMENTS AND REPORTS

In the event of serious announcements, they will be performed according to Art. 21 (HFV).

PUBLICATION AND DISSEMINATION POLICY

Publication of results

Publication of the study results is planned. An acknowledgement to the Clinical Trials Unit (CTU) St. Gallen is enclosed in any publication that will result from this study. The study will be registered at clinicaltrials.gov.

FUNDING AND SUPPORT

No funding necessary.

INSURANCE

In the event of study-related damage or injuries, the public liability insurance of the Sponsor (i.e. the Kantonsspital St. Gallen) provides compensation, except for claims that arise from wilful misconduct or gross negligence.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Low grade glioma, cavernoma, metastasis
* age ≥ 18 years < 65 years

Exclusion Criteria:

* No given operability for anaesthetic reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive ongoing recruitment through investigator(s) in daily clinical practice (consultations). The subjects will receive the consent form with an address and phone number indicated where further questions regarding the study can be discussed directly with the project leader. This will take place at least one week before the hospitalisation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Changes in Pain and Anxiety (NRS) | 1st day preop, intraoperatively, 3rd day postop, 6th month postop
  Numeric rating scale (NRS). (Kremer et al., 1981; Farrar et al., 2000) Preoperative assessment of anxiety is evaluated using the NRS on a scale of 0-10. Intraoperatively the NRS is used at three time points to assess for anxiety and pain. 0 indicates the absence of pain or anxiety, whereas 10 indicates the maximum possible patients' perception of pain or anxiety

SECONDARY OUTCOMES:
Cognition | 1st preoperative day
  Mini-Mental State Examination (MMSE, Folstein et al., 1983)
Changes in General psychological symptoms | 1st preoperative day, 3rd day postoperative visit, 6th month postop
  The patients health questionnaire (PHQ-D, Gräfe et al., 2004)
Changes in General psychological symptoms | 1st preoperative day, 6th month postop
  Beck Depression Inventory (BDI, Beck et al., 1961)
Changes in Stress and Anxiety | 1st preoperative day, 3rd day postoperative visit, 6th month postop
  The Hospital Anxiety and Depression Scale (HADS-D, Bjelland et al., 2002)
Changes in Stress and Anxiety | 1st preoperative day, 3rd day postoperative visit, 6th month postop
  The Posttraumatic Stress Diagnostic Scale (PDS-1, Griesel et al., 2006)
Changes in Pain | 1st preoperative day, 3rd day postoperative visit, 6th month postop
  The Brief Pain Inventory (BPI, Cleeland and Ryan, 1994; Radbruch et al., 1999)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Surbeck, MD, Principal Investigator — Department of Neurosurgery, Cantonal Hospital St. Gallen, Switzerland
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, St.Gallen, Switzerland

REFERENCES:
- [Background] Verordnung über die Humanforschung mit Ausnahme der klinischen Versuche (Humanforschungsverordnung, HFV) / Ordonnance relative à la recherche sur l'être humain à l'exception des essais cliniques (Ordonnance relative à la recherche sur l'être humain, ORH) / Ordinance on Human Research with the Exception of Clinical Trials (Human Research Ordinance, HRO)
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. PLoS Med. 2007 Oct 16;4(10):e296. doi: 10.1371/journal.pmed.0040296. PMID 17941714
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. PLoS Med. 2007 Oct 16;4(10):e297. doi: 10.1371/journal.pmed.0040297. PMID 17941715
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Farrar JT, Portenoy RK, Berlin JA, Kinman JL, Strom BL. Defining the clinically important difference in pain outcome measures. Pain. 2000 Dec 1;88(3):287-294. doi: 10.1016/S0304-3959(00)00339-0. PMID 11068116
- [Background] Folstein MF, Robins LN, Helzer JE. The Mini-Mental State Examination. Arch Gen Psychiatry. 1983 Jul;40(7):812. doi: 10.1001/archpsyc.1983.01790060110016. No abstract available. PMID 6860082
- [Background] Griesel D, Wessa M, Flor H. Psychometric qualities of the German version of the Posttraumatic Diagnostic Scale (PTDS). Psychol Assess. 2006 Sep;18(3):262-8. doi: 10.1037/1040-3590.18.3.262. PMID 16953729
- [Background] Gräfe K, Zipfel S, Herzog W, Löwe B. Screening psychischer Störungen mit dem "Gesundheitsfragebogen für Patienten (PHQ-D)" Daignostica 2004; 50(4): 11
- [Background] Keefe FJ, Lumley M, Anderson T, Lynch T, Studts JL, Carson KL. Pain and emotion: new research directions. J Clin Psychol. 2001 Apr;57(4):587-607. doi: 10.1002/jclp.1030. PMID 11255208
- [Background] Kremer E, Atkinson HJ, Ignelzi RJ. Measurement of pain: patient preference does not confound pain measurement. Pain. 1981 Apr;10(2):241-248. doi: 10.1016/0304-3959(81)90199-8. PMID 7267140
- [Background] Milian M, Tatagiba M, Feigl GC. Patient response to awake craniotomy - a summary overview. Acta Neurochir (Wien). 2014 Jun;156(6):1063-70. doi: 10.1007/s00701-014-2038-4. Epub 2014 Mar 5. PMID 24595540
- [Background] Radbruch L, Loick G, Kiencke P, Lindena G, Sabatowski R, Grond S, Lehmann KA, Cleeland CS. Validation of the German version of the Brief Pain Inventory. J Pain Symptom Manage. 1999 Sep;18(3):180-7. doi: 10.1016/s0885-3924(99)00064-0. PMID 10517039
- See also: Declaration of Helsinki, Version November 2013 — https://www.wma.net/wp-content/uploads/2016/11/DoH-Oct2013-JAMA.pdf
- See also: Essentials of Good Epidemiological Practice — https://public-health.ch/documents/91/EGEP_en.pdf
- See also: Human Research Act, Federal Law about Research involving Human Subjects — https://www.admin.ch/opc/en/classified-compilation/20061313/201401010000/810.30.pdf